CLINICAL TRIAL: NCT02414477
Title: Metabolism of Deuterated NNN in Smokeless Tobacco Users
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: not successful in securing the deuterated products
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014NTLS110
Record Dates: First submitted 2015-03-23; First posted 2015-04-10 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Toxicant Exposure
Keywords: tobacco toxicants; smokeless tobacco; nitrosamines; tobacco specific nitrosamines (TSNAs)
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smokeless tobacco study product (Experimental): Smokeless tobacco product spiked with deuterated NNN.
  Interventions: Drug: Deuterated NNN

INTERVENTIONS:
Drug: Deuterated NNN — Smokeless tobacco study product

SUMMARY:
The purpose of this study is to better understand how people break down a tobacco specific cancer-causing toxin called N'-nitrosonornicotine (NNN) that is present in smokeless tobacco and cigarettes. Some people are able to get rid of this chemical as a harmless agent better than others. Through this research, the investigators hope to develop a better understanding of how people process potentially harmful chemicals and identify tobacco users who are in danger of developing cancer. Participants will complete questionnaires regarding their health and smoking history. The investigators will take blood samples, saliva samples, cheek cells and urine to measure exposure to toxins and harmful chemicals present in smokeless tobacco. Participants will be given smokeless tobacco study product and be asked to use only it for the entire time they are in the study. The study product contains deuterated NNN. Deuterated NNN is just like the NNN found in commercially available smokeless tobacco products, but is labeled with deuterium or heavy hydrogen atoms. Deuterium is non-toxic and safe. Using smokeless tobacco containing deuterium allows us to follow NNN as it is broken down in the body.

DETAILED DESCRIPTION:
Fifty healthy smokeless tobacco users will be recruited by advertising in Minneapolis-St. Paul area. This research will be conducted at the Tobacco Research Center at the University of Minnesota. Regular smokeless tobacco users will be screened over the phone. If eligible after the phone screen, participants will be invited to attend an orientation visit in the clinic where consent will be obtained and subjects will fill out forms about their tobacco use and medical history. Subjects who are determined to be eligible after the orientation visit will return to the clinic for a baseline visit where they will receive the smokeless tobacco product and be instructed to use only the study product until they return for their first lab session seven days later.

Prior to each of the three lab sessions, subjects will collect all of their urine for the 24 hours leading up to their scheduled appointment. At each lab session, participants will use the study product and collect their saliva and tobacco juices at regular intervals. Participants will also swab the inside of their cheek for cells and have their blood drawn.

Collected samples will be used to characterize the metabolic activation and DNA binding of NNN.

ELIGIBILITY:
Inclusion Criteria:

* Regular smokeless tobacco user
* Good physical health with no unstable medical conditions
* Stable and good mental health, i.e., currently do not experience unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria, during the past six months
* Willing to perform study activities such as having blood sample drawn, saliva collection, urine collection, multiple clinic visits
* For female subjects of child bearing potential, not known to be pregnant or nursing, or planning to become pregnant within next 12 months
* Provide written informed consent

Exclusion Criteria:

* Using other tobacco or nicotine containing products
* Unstable medical condition
* Currently taking any medications that affect relevant metabolic enzymes
* Not willing to use switch smokeless tobacco brand to use tobacco enriched with [pyridine-D4](S)-NNN for the course of this study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Determine extent of α-hydroxylation of NNN as indicated by presence of keto acid 17 and hydroxy acid 22 in plasma | One week post dosing
  Deuterated NNN will be assessed after one week of regular use via smokeless tobacco study product, as well as during use in three lab sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Boyle, P. and Levin, P. (2008) World Cancer Report, 2008. IARC, Lyon, FR.
- [Background] World Health Organization. (2012) Cancer Fact Sheet No. 297, February 2012 (http://www.who.int/mediacentre/factsheets/fs297/en/index.html).
- [Background] Fontham ET, Thun MJ, Ward E, Portier KM, Balch AJ, Delancey JO, Samet JM; ACS Cancer and the Environment Subcommittee. American Cancer Society perspectives on environmental factors and cancer. CA Cancer J Clin. 2009 Nov-Dec;59(6):343-51. doi: 10.3322/caac.20041. Epub 2009 Oct 28. PMID 19864396
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Personal habits and indoor combustions. IARC Monogr Eval Carcinog Risks Hum. 2012;100(Pt E):1-538. No abstract available. PMID 23193840
- [Background] Centers for Disease Control and Prevention (CDC). Current cigarette smoking among adults - United States, 2011. MMWR Morb Mortal Wkly Rep. 2012 Nov 9;61(44):889-94. PMID 23134971
- [Background] Shafey, O., Eriksen, M.P., Ross, H., and Mackay, J. (2009) The Tobacco Atlas, 3rd Edition. American Cancer Society and World Lung Foundation, Atlanta, GA.
- [Background] United States Department of Health and Human Services (2009) National Survey on Drug Use and Health. Department of Health and Human Services, Substance Abuse and Mental Health Services Administration, Office of Applied Studies, Washington, D.C.
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Smokeless tobacco and some tobacco-specific N-nitrosamines. IARC Monogr Eval Carcinog Risks Hum. 2007;89:1-592. No abstract available. PMID 18335640
- [Background] Fiore, M.C., Jaén, C.R., and Baker, T.B. (2008) Treating Tobacco Use and Dependence: 2008 Update. Clinical Practice Guideline. U.S. Department of Health and Human Services. Public Health Service., Rockville, MD.
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Institute of Medicine (2012) Scientific Standards for Studies on Modified Risk Tobacco Products. National Academy Press, Washington, D.C.
- [Background] Surveillance Research Program, N. C. I. (2013) Fast Stats: An interactive tool for access to SEER cancer statistics. http://seer.cancer.gov/faststats (Accessed on 5-21-2013).
- [Background] American Nonsmokers' Rights Foundation. (2013) Percent of Population Covered by 100% Smokefree Restaurant AND Bar Laws. http://no-smoke.org/pdf/RBpercentMap. pdf .
- [Background] Centers for Disease Control and Prevention (US); National Center for Chronic Disease Prevention and Health Promotion (US); Office on Smoking and Health (US). How Tobacco Smoke Causes Disease: The Biology and Behavioral Basis for Smoking-Attributable Disease: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK53017/ PMID 21452462
- [Background] Hecht SS. Tobacco smoke carcinogens and lung cancer. J Natl Cancer Inst. 1999 Jul 21;91(14):1194-210. doi: 10.1093/jnci/91.14.1194. PMID 10413421
- [Background] Greenman, C., Stephens, P., Smith, R., Dalgliesh, G. L., Hunter, C., Bignell, G., Davies, H., Teague, J., Butler, A., Stevens, C., Edkins, S., O'Meara, S., Vastrik, I., Schmidt, E. E., Avis, T., Barthorpe, S., Bhamra, G., Buck, G., Choudhury, B., Clements, J., Cole, J., Dicks, E., Forbes, S., Gray, K., Halliday, K., Harrison, R., Hills, K., Hinton, J., Jenkinson, A., Jones, D., Menzies, A., Mironenko, T., Perry, J., Raine, K., Richardson, D., Shepherd, R., Small, A., Tofts, C., Varian, J., Webb, T., West, S., Widaa, S., Yates, A., Cahill, D. P., Louis, D. N., Goldstraw, P., Nicholson, A. G., Brasseur, F., Looijenga, L., Weber, B. L., Chiew, Y. E., DeFazio, A., Greaves, M. F., Green, A. R., Campbell, P., Birney, E., Easton, D. F., Chenevix-Trench, G., Tan, M. H., Khoo, S. K., Teh, B. T., Yuen, S. T., Leung, S. Y., Wooster, R., Futreal, P. A., and Stratton, M. R. (2007) Patterns of somatic mutation in human cancer genomes. Nature 446, 153-158.
- [Background] Ding, L., Getz, G., Wheeler, D. A., Mardis, E. R., McLellan, M. D., Cibulskis, K., Sougnez, C., Greulich, H., Muzny, D. M., Morgan, M. B., Fulton, L., Fulton, R. S., Zhang, Q., Wendl, M. C., Lawrence, M. S., Larson, D. E., Chen, K., Dooling, D. J., Sabo, A., Hawes, A. C., Shen, H., Jhangiani, S. N., Lewis, L. R., Hall, O., Zhu, Y., Mathew, T., Ren, Y., Yao, J., Scherer, S. E., Clerc, K., Metcalf, G. A., Ng, B., Milosavljevic, A., Gonzalez-Garay, M. L., Osborne, J. R., Meyer, R., Shi, X., Tang, Y., Koboldt, D. C., Lin, L., Abbott, R., Miner, T. L., Pohl, C., Fewell, G., Haipek, C., Schmidt, H., Dunford-Shore, B. H., Kraja, A., Crosby, S. D., Sawyer, C. S., Vickery, T., Sander, S., Robinson, J., Winckler, W., Baldwin, J., Chirieac, L. R., Dutt, A., Fennell, T., Hanna, M., Johnson, B. E., Onofrio, R. C., Thomas, R. K., Tonon, G., Weir, B. A., Zhao, X., Ziaugra, L., Zody, M. C., Giordano, T., Orringer, M. B., Roth, J. A., Spitz, M. R., Wistuba, I. I., Ozenberger, B., Good, P. J., Chang, A. C., Beer, D. G., Watson, M. A., Ladanyi, M., Broderick, S., Yoshizawa, A., Travis, W. D., Pao, W., Province, M. A., Weinstock, G. M., Varmus, H. E., Gabriel, S. B., Lander, E. S., Gibbs, R. A., Meyerson, M., and Wilson, R. K. (2008) Somatic mutations affect key pathways in lung adenocarcinoma. Nature 455, 1069-1075.
- [Background] Pleasance ED, Stephens PJ, O'Meara S, McBride DJ, Meynert A, Jones D, Lin ML, Beare D, Lau KW, Greenman C, Varela I, Nik-Zainal S, Davies HR, Ordonez GR, Mudie LJ, Latimer C, Edkins S, Stebbings L, Chen L, Jia M, Leroy C, Marshall J, Menzies A, Butler A, Teague JW, Mangion J, Sun YA, McLaughlin SF, Peckham HE, Tsung EF, Costa GL, Lee CC, Minna JD, Gazdar A, Birney E, Rhodes MD, McKernan KJ, Stratton MR, Futreal PA, Campbell PJ. A small-cell lung cancer genome with complex signatures of tobacco exposure. Nature. 2010 Jan 14;463(7278):184-90. doi: 10.1038/nature08629. Epub 2009 Dec 16. PMID 20016488
- [Background] Lee W, Jiang Z, Liu J, Haverty PM, Guan Y, Stinson J, Yue P, Zhang Y, Pant KP, Bhatt D, Ha C, Johnson S, Kennemer MI, Mohan S, Nazarenko I, Watanabe C, Sparks AB, Shames DS, Gentleman R, de Sauvage FJ, Stern H, Pandita A, Ballinger DG, Drmanac R, Modrusan Z, Seshagiri S, Zhang Z. The mutation spectrum revealed by paired genome sequences from a lung cancer patient. Nature. 2010 May 27;465(7297):473-7. doi: 10.1038/nature09004. PMID 20505728
- [Background] Pfeifer GP, Denissenko MF, Olivier M, Tretyakova N, Hecht SS, Hainaut P. Tobacco smoke carcinogens, DNA damage and p53 mutations in smoking-associated cancers. Oncogene. 2002 Oct 21;21(48):7435-51. doi: 10.1038/sj.onc.1205803. PMID 12379884
- [Background] Govindan R, Ding L, Griffith M, Subramanian J, Dees ND, Kanchi KL, Maher CA, Fulton R, Fulton L, Wallis J, Chen K, Walker J, McDonald S, Bose R, Ornitz D, Xiong D, You M, Dooling DJ, Watson M, Mardis ER, Wilson RK. Genomic landscape of non-small cell lung cancer in smokers and never-smokers. Cell. 2012 Sep 14;150(6):1121-34. doi: 10.1016/j.cell.2012.08.024. PMID 22980976
- [Background] Vogelstein B, Papadopoulos N, Velculescu VE, Zhou S, Diaz LA Jr, Kinzler KW. Cancer genome landscapes. Science. 2013 Mar 29;339(6127):1546-58. doi: 10.1126/science.1235122. PMID 23539594
- [Background] Burns DM, Dybing E, Gray N, Hecht S, Anderson C, Sanner T, O'Connor R, Djordjevic M, Dresler C, Hainaut P, Jarvis M, Opperhuizen A, Straif K. Mandated lowering of toxicants in cigarette smoke: a description of the World Health Organization TobReg proposal. Tob Control. 2008 Apr;17(2):132-41. doi: 10.1136/tc.2007.024158. No abstract available. PMID 18375736
- [Background] U.S.Food and Drug Administration (2012) Harmful and Potentially Harmful Constituents in Tobacco Products and Tobacco Smoke; Established List. Fed. Regist. 77, 20034-20037.
- [Background] Hecht SS. Biochemistry, biology, and carcinogenicity of tobacco-specific N-nitrosamines. Chem Res Toxicol. 1998 Jun;11(6):559-603. doi: 10.1021/tx980005y. No abstract available. PMID 9625726
- [Background] U.S.Department of Health and Human Services. (2013) National Toxicology Program. http://ntp.niehs.nih.gov/
- [Background] Vogel RI, Carmella SG, Stepanov I, Hatsukami DK, Hecht SS. The ratio of a urinary tobacco-specific lung carcinogen metabolite to cotinine is significantly higher in passive than in active smokers. Biomarkers. 2011 Sep;16(6):491-7. doi: 10.3109/1354750X.2011.598565. Epub 2011 Aug 3. PMID 21812592
- [Background] Hecht SS. Tobacco carcinogens, their biomarkers and tobacco-induced cancer. Nat Rev Cancer. 2003 Oct;3(10):733-44. doi: 10.1038/nrc1190. PMID 14570033
- [Background] Yuan JM, Gao YT, Murphy SE, Carmella SG, Wang R, Zhong Y, Moy KA, Davis AB, Tao L, Chen M, Han S, Nelson HH, Yu MC, Hecht SS. Urinary levels of cigarette smoke constituent metabolites are prospectively associated with lung cancer development in smokers. Cancer Res. 2011 Nov 1;71(21):6749-57. doi: 10.1158/0008-5472.CAN-11-0209. Epub 2011 Oct 25. PMID 22028322
- [Background] Yuan JM, Knezevich AD, Wang R, Gao YT, Hecht SS, Stepanov I. Urinary levels of the tobacco-specific carcinogen N'-nitrosonornicotine and its glucuronide are strongly associated with esophageal cancer risk in smokers. Carcinogenesis. 2011 Sep;32(9):1366-71. doi: 10.1093/carcin/bgr125. Epub 2011 Jul 6. PMID 21734256
- [Background] Hecht SS, Chen CB, Ornaf RM, Jacobs E, Adams JD, Hoffmann D. Reaction of nicotine and sodium nitrite: formation of nitrosamines and fragmentation of the pyrrolidine ring. J Org Chem. 1978 Jan 6;43(1):72-6. doi: 10.1021/jo00395a017. No abstract available. PMID 619049
- [Background] Hecht SS, Chen CB, Hirota N, Ornaf RM, Tso TC, Hoffmann D. Tobacco-specific nitrosamines: formation from nicotine in vitro and during tobacco curing and carcinogenicity in strain A mice. J Natl Cancer Inst. 1978 Apr;60(4):819-24. doi: 10.1093/jnci/60.4.819. PMID 633391
- [Background] Hecht SS, Carmella SG, Murphy SE, Akerkar S, Brunnemann KD, Hoffmann D. A tobacco-specific lung carcinogen in the urine of men exposed to cigarette smoke. N Engl J Med. 1993 Nov 18;329(21):1543-6. doi: 10.1056/NEJM199311183292105. PMID 8413477
- [Background] Carmella SG, Akerkar S, Hecht SS. Metabolites of the tobacco-specific nitrosamine 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone in smokers' urine. Cancer Res. 1993 Feb 15;53(4):721-4. PMID 8428352
- [Background] Singer, B. and Grunberger, D. (1983) Molecular Biology of Mutagens and Carcinogens. Plenum Press, New York.
- [Background] Haglund J, Rafiq A, Ehrenberg L, Golding BT, Tornqvist M. Transalkylation of phosphotriesters using Cob(I)alamin: toward specific determination of DNA-phosphate adducts. Chem Res Toxicol. 2000 Apr;13(4):253-6. doi: 10.1021/tx990135m. PMID 10775324
- [Background] Reynolds M, Peterson E, Quievryn G, Zhitkovich A. Human nucleotide excision repair efficiently removes chromium-DNA phosphate adducts and protects cells against chromate toxicity. J Biol Chem. 2004 Jul 16;279(29):30419-24. doi: 10.1074/jbc.M402486200. Epub 2004 Apr 15. PMID 15087443
- [Background] Haglund J, Van Dongen W, Lemiere F, Esmans EL. Analysis of DNA-phosphate adducts in vitro using miniaturized LC-ESI-MS/MS and column switching: phosphotriesters and alkyl cobalamins. J Am Soc Mass Spectrom. 2004 Apr;15(4):593-606. doi: 10.1016/j.jasms.2003.12.012. PMID 15047064
- [Background] Beranek DT, Weis CC, Swenson DH. A comprehensive quantitative analysis of methylated and ethylated DNA using high pressure liquid chromatography. Carcinogenesis. 1980 Jul;1(7):595-606. doi: 10.1093/carcin/1.7.595. PMID 11219835
- [Background] Haglund J, Henderson AP, Golding BT, Tornqvist M. Evidence for phosphate adducts in DNA from mice treated with 4-(N-Methyl-N-nitrosamino)-1-(3-pyridyl)-1-butanone (NNK). Chem Res Toxicol. 2002 Jun;15(6):773-9. doi: 10.1021/tx015542o. PMID 12067244
- [Background] Zhang S, Wang M, Villalta PW, Lindgren BR, Lao Y, Hecht SS. Quantitation of pyridyloxobutyl DNA adducts in nasal and oral mucosa of rats treated chronically with enantiomers of N'-nitrosonornicotine. Chem Res Toxicol. 2009 May;22(5):949-56. doi: 10.1021/tx900040j. PMID 19405515
- [Background] Zhang S, Wang M, Villalta PW, Lindgren BR, Upadhyaya P, Lao Y, Hecht SS. Analysis of pyridyloxobutyl and pyridylhydroxybutyl DNA adducts in extrahepatic tissues of F344 rats treated chronically with 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone and enantiomers of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol. Chem Res Toxicol. 2009 May;22(5):926-36. doi: 10.1021/tx900015d. PMID 19358518
- [Background] Lao Y, Yu N, Kassie F, Villalta PW, Hecht SS. Analysis of pyridyloxobutyl DNA adducts in F344 rats chronically treated with (R)- and (S)-N'-nitrosonornicotine. Chem Res Toxicol. 2007 Feb;20(2):246-56. doi: 10.1021/tx060208j. PMID 17305408